CLINICAL TRIAL: NCT02036866
Title: Corticospinal Excitability and Rehab in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-16794
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; grade I and II knee osteoarthritis; arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Lymphoma, Follicular; Arthritis | interventions — Transcutaneous Electric Nerve Stimulation; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physical Therapy Positive Expectation (Experimental): The physical therapist will read a script indicating that the intervention is an effective treatment for knee osteoarthritis and is expected to reduce pain and improve strength. Patients are then instructed on the home exercise program and how to operate the TENS (transcutaneous electrical nerve stimulation) unit. The duration of intervention is 1 week during which patients will wear then wear the TENS unit for 8 hours per day and perform no more than 3 sets of 10 repetitions of the physical therapy exercises daily.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation; Other: Physical Therapy Exercises
- Physical Therapy Neutral Expectation (Experimental): The physical therapist will read a script indicating that the intervention may or may not be an effective treatment for knee osteoarthritis and may nor may not reduce pain and improve strength. Patients are then instructed on the home exercise program and how to operate the TENS unit. The duration of intervention is 1 week during which patients will wear then wear the TENS unit for 8 hours per day and perform no more than 3 sets of 10 repetitions of the physical therapy exercises daily.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation; Other: Physical Therapy Exercises
- Control- No Intervention (Experimental): The patients in the control group will be reminded of their appointment in 1 week and instructed to maintain their usual activity level during that time.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulation — The TENS electrodes will be applied on the medial and lateral superior, as well as the medial and lateral inferior, borders of the patella. A continuous biphasic pulsatile current (150 Hz, phase duration 150 µs) will be applied at an intensity that produces a comfortable sensation but not a muscle contraction. The duration of intervention will be 8 hours per day for 1 week.
  Other Names: TENS; Sensory TENS
  Arms: Physical Therapy Neutral Expectation; Physical Therapy Positive Expectation
Other: Physical Therapy Exercises — Patients will be given detailed verbal and hands-on instruction in a home exercise program. This program will consist of 6 exercises modeled from established protocols focuses on improving lower extremity strength. Patients will be instructed to do the exercises daily and to progress the exercises over the week for a maximum of 30 repetitions per day for 1 week.
  Arms: Physical Therapy Neutral Expectation; Physical Therapy Positive Expectation
Other: No Intervention — Patients will be instructed to maintain their usual activity level.
  Arms: Control- No Intervention

SUMMARY:
To determine differences in thigh muscle function in individuals with and without knee arthritis, and also determine the effectiveness of common physical therapy interventions on clinical and patient oriented outcomes.

DETAILED DESCRIPTION:
The primary objective of the proposed research evaluates the concurrent changes in corticospinal excitability and central sensitization of pain pathways for their influence on quadriceps voluntary activation. A secondary objective is to establish the feasibility of an intervention study to determine if changes in the excitability of these supraspinal motor and sensory processes can be modified by physical therapy interventions targeting pain and muscle strengthening. We hypothesize that patients with knee osteoarthritis will show measurable deficits in quadriceps voluntary activation that can be explained by lower levels of corticospinal excitability and increased pain sensitization. A 1 week physical therapy intervention will improve voluntary activation and reduce pain with concurrent changes in underlying motor and sensory processes. We further hypothesize that part of this improvement will be attributed to positive treatment expectation.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-65
* Grade I or II knee Osteoarthritis confirmed by radiographs or other imaging and at least one of the following:

  * Age > 50 years old
  * Morning stiffness < 30 minutes
  * Crepitus
* Meet at least 3 of 6 diagnostic criteria for osteoarthritis:

  * Age > 50 years old
  * Morning stiffness < 30 minutes
  * Crepitus
  * Bony tenderness
  * Bony enlargement
  * No palpable warmth

Exclusion Criteria:

* BMI > 30
* History of traumatic spine or lower extremity injury within the last 6 months
* Previous adverse reaction to electrical stimulation (i.e. burns or hypersensitivity)
* Cardiac pacemaker
* Metal implants in head
* Current pregnancy
* Neurological disorders
* History of seizures
* Unable to give consent or understand the procedures of this study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in quadriceps force output and voluntary activation | Baseline and following 1 week intervention (2 Study Visits)
  Quadriceps activation will be estimated by utilizing the burst-superimposition technique on a maximum voluntary isometric contraction (MVIC) and during a resting condition. The burst-superimposition technique provides the muscle with a percutaneous stimulus to recruit any remaining muscle fibers which have not been stimulated.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Grindstaff, PhD, PT, ATC, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States